CLINICAL TRIAL: NCT00794300
Title: Reproducibility of Myocardial Salvage Index in Acute Myocardial Infarction by Cardiac Magnetic Resonance Imaging
Brief Title: Reproducibility of Magnetic Resonance Myocardial Salvage Index
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Holger Thiele, Director, University of Leipzig
Other Study IDs: Repro100
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Myocardial Infarction
Keywords: reproducibility; contrast agent; magnetic resonance imaging; infarct size; myocardial salvage index; myocardial salvage assessment
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute myocardial infarction patients
  Interventions: Device: second magnetic resonance imaging scan

INTERVENTIONS:
Device: second magnetic resonance imaging scan

SUMMARY:
The myocardial salvage assessed by using multimodal cardiac magnetic resonance imaging is a rather new technique which can be used as a surrogate endpoint to reduce the sample size in studies comparing different reperfusion strategies in myocardial infarction. As reproducibility of myocardial salvage has not been evaluated appropriately, we aim to scan 20 patients on 2 subsequent days to evaluate reproducibility of myocardial salvage index.

ELIGIBILITY:
Inclusion Criteria:

* ST-elevation myocardial infarction
* Primary percutaneous coronary intervention

Exclusion Criteria:

* Contraindications for magnetic resonance imaging

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ST-elevation myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2008-11-01 (Actual); Primary Completion 2009-11-01 (Actual); Study Completion 2010-05-01 (Actual)

PRIMARY OUTCOMES:
Myocardial salvage index reproducibility | 2 days

SECONDARY OUTCOMES:
infarct size reproducibility | 2 days
area at risk reproducibility | 2 days
microvascular obstruction reproducibility | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (1):
- University of Leipzig - Heart Center, Leipzig, Germany

REFERENCES:
- [Derived] Desch S, Engelhardt H, Meissner J, Eitel I, Sareban M, Fuernau G, de Waha S, Grothoff M, Gutberlet M, Schuler G, Thiele H. Reliability of myocardial salvage assessment by cardiac magnetic resonance imaging in acute reperfused myocardial infarction. Int J Cardiovasc Imaging. 2012 Feb;28(2):263-72. doi: 10.1007/s10554-011-9802-9. Epub 2011 Jan 30. PMID 21279689